CLINICAL TRIAL: NCT05122208
Title: Clinical Effects of Famotidine Use in Intensive Care Covid-19 Patients
Brief Title: Famotidine in Covid-19 Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: istanbulMU intensive care
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 Intensive Care Unit; Famotidine; mortality; entubation
MeSH Terms: conditions — COVID-19 | interventions — Famotidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Famotidine Group: Patients who were administered Famotidine 160 mg/day PO or nasogastric.
  Interventions: Drug: Famotidine Tablets
- Control Group: Patients who were not administered Famotidine

INTERVENTIONS:
Drug: Famotidine Tablets — 160 mg/day Famotidine
  Groups: Famotidine Group

SUMMARY:
The COVID-19 disease, caused by SARS-CoV-2 virus, started in December 2019 and created a pandemic with high mortality and morbidity. Since a fully proven treatment has not been developed, the efficacy of currently available treatments is being investigated. Famotidine, an H2Receptor blocker, is one of the drug treatments being investigated. In this study, we aimed to investigate the effect of Famotidine treatment on the clinic and mortality of Covid-19 patients treated in the intensive care unit.

DETAILED DESCRIPTION:
The computer and written records of the patients followed in the Covid-19 Intensive Care Units of a research hospital during the pandemic process will be examined. Patients over the age of 18 who have SARS-CoV-2 mRNA detected by nasopharyngeal PCR (Polymeraze Chaine Reaction) will be included in the study. Patients with immunosuppression, end-stage renal disease, liver disease, G6PD deficiency, ALT/AST >5, long QT syndrome in ECG, diagnosed with psoriasis, porphyria, pregnant, and allergic reactions to famotidine or similar drugs were excluded from the study. Patients' age, gender, comorbidities, smoking and APACHE II score will be recorded. Patients who were administered Famotidine 160 mg/day PO or nasogastric and were not given this treatment since their admission to the intensive care unit will be compared. The primary outcome will be the need for invasive mechanical ventilation, intensive care mortality, and both. As a secondary outcome, serum markers indicating the severity of the disease (Leukocytes, lymphocytes, neutrophils/leukocytes, platelets, ferritin, CRP, D-Dimer, fibrinogen, procalcitonin, IL-6, troponin, creatinine, AST, ALT, P/F ratio and lactate) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have SARS-CoV-2 mRNA detected by nasopharyngeal PCR

Exclusion Criteria:

* immunosuppression
* end-stage renal disease
* liver disease
* G6PD deficiency
* long QT syndrome in ECG
* psoriasis
* porphyria
* pregnant
* allergic reactions to famotidine or similar drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients followed in the Covid-19 Intensive Care Units
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Number of patients who died in intensive care | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  Mortality in intensive care
Number of patients who were intubated in intensive care | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  Development of respiratory distress requiring intubation in the patient

SECONDARY OUTCOMES:
Ferritin | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  Ferritin in nonogram/miiliter
CRP | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  C-Reactive protein in miligram/liter
D-Dimer | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  D-Dimer in nonogram/miiliter
Fibrinogen | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  Fibrinogen in nonogram/miiliter
Procalcitonin | Within 17 days from the patient's admission to the intensive care unit or if he dies within this period, to this date
  Procalcitonin in nonogram/miiliter

CONTACTS AND LOCATIONS:
Overall Officials: mesure Gul Nihan Ozden, MD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided